CLINICAL TRIAL: NCT04458857
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing the Efficacy, Safety, and Tolerability of Subcutaneous Administration of Fremanezumab Versus Placebo for the Preventive Treatment of Episodic Migraine in Pediatric Patients 6 to 17 Years of Age
Brief Title: A Study to Test if Fremanezumab is Effective in Preventing Episodic Migraine in Patients 6 to 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-CNS-30083; 2019-002055-42 (EudraCT Number)
Record Dates: First submitted 2020-06-22; First posted 2020-07-07 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Migraine
Keywords: episodic migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fremanezumab Dose A (Experimental): Participants weighing <threshold weight will receive fremanezumab SC at dose A for 3 months.
  Interventions: Drug: Fremanezumab
- Fremanezumab Dose B (Experimental): Participants weighing ≥threshold weight will receive fremanezumab SC at dose B for 3 months.
  Interventions: Drug: Fremanezumab
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Dose A or Dose B subcutaneous
  Arms: Fremanezumab Dose A; Fremanezumab Dose B
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of fremanezumab as compared to placebo for the preventive treatment of episodic migraine (EM).

Secondary objectives are to further demonstrate the efficacy of fremanezumab as compared to placebo for the preventive treatment of EM, to evaluate the safety and tolerability of fremanezumab in the preventive treatment of EM and to evaluate the immunogenicity of fremanezumab and the impact of antidrug antibodies (ADAs) on clinical outcomes in participants exposed to fremanezumab.

The total duration of the study is planned to be up to 51 months.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a clinical history of recurrent headache consistent with the diagnosis of migraine for at least 6 months before screening, consistent with ICHD-3 criteria (Headache Classification Committee of the IHS 2013), and a history of ≤=14 headache days per month in each of the 3 months prior to screening (visit 1).
* The participant or parent/caregiver maintain a prospectively collected headache diary
* The participant does not have chronic daily headache. For the purposes of this study, chronic daily headache is operationally defined as <4 headache-free days during the 28-day baseline period.

NOTE: Additional criteria apply; please contact the investigator for more information.

Exclusion Criteria:

* The participant is using medications containing opioids (including codeine) or barbiturates (including Fiorinal®, Fioricet®, or any other combination containing butalbital) for the treatment of migraine during the 3 months prior to the day of the screening visit.
* The participant or parent/caregiver maintain a prospectively collected headache diary
* The participant has used an intervention/device (eg, scheduled nerve block or transcranial magnetic stimulation) for the treatment of migraine or in the head or neck area for any condition during the 2 months prior to the day of the screening visit.
* The participant has a current history of a clinically significant psychiatric condition, at the discretion of the investigator. Any prior history of a suicide attempt, or a history of suicidal ideation with a specific plan within the past 2 years, must be excluded.
* The participant has an ongoing infection or a known history of human immunodeficiency virus infection, tuberculosis, Lyme disease, or chronic hepatitis B or C, or a known active infection of coronavirus disease 2019 (COVID-19).
* The participant has a past or current history of cancer.
* The participant is pregnant or nursing.
* The participant has a history of hypersensitivity reactions to injected proteins, including mAbs, or a history of Stevens-Johnson Syndrome or toxic epidermal necrolysis syndrome, or the participant is concomitantly using lamotrigine.
* The participant received a live attenuated vaccine (eg, intranasal flu vaccine, and measles, mumps, and rubella vaccine) within the 12-week period prior to screening. Note: If a medical need arises during the study, the participant may receive a live attenuated vaccine.
* The participant has a current or past medical history of hemiplegic migraine.

NOTE: Additional criteria apply; please contact the investigator for more information.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (89):
- United States (45):
  - Teva Investigational Site 14281, Little Rock, Arkansas
  - Teva Investigational Site 14253, Banning, California
  - Teva Investigational Site 14370, Loma Linda, California
  - Teva Investigational Site 14322, Los Angeles, California
  - Teva Investigational Site 14361, Sacramento, California
  - Teva Investigational Site 14319, Aurora, Colorado
  - Teva Investigational Site 14368, Colorado Springs, Colorado
  - Teva Investigational Site 14244, Jacksonville, Florida
  - Teva Investigational Site 14325, Miami, Florida
  - Teva Investigational Site 14250, West Palm Beach, Florida
  - Teva Investigational Site 14255, West Palm Beach, Florida
  - Teva Investigational Site 14243, Atlanta, Georgia
  - Teva Investigational Site 14258, Savannah, Georgia
  - Teva Investigational Site 14263, Hoffman Estates, Illinois
  - Teva Investigational Site 14283, Park Ridge, Illinois
  - Teva Investigational Site 14245, Wichita, Kansas
  - Teva Investigational Site 14327, Louisville, Kentucky
  - Teva Investigational Site 14360, Covington, Louisiana
  - Teva Investigational Site 14365, Baltimore, Maryland
  - Teva Investigational Site 14317, Silver Spring, Maryland
  - Teva Investigational Site 14246, Waltham, Massachusetts
  - Teva Investigational Site 14251, Ann Arbor, Michigan
  - Teva Investigational Site 14270, Minneapolis, Minnesota
  - Teva Investigational Site 14376, Ridgeland, Mississippi
  - Teva Investigational Site 14256, Bridgeton, Missouri
  - Teva Investigational Site 14371, New Brunswick, New Jersey
  - Teva Investigational Site 14276, Amherst, New York
  - Teva Investigational Site 14377, Durham, North Carolina
  - Teva Investigational Site 14248, Raleigh, North Carolina
  - Teva Investigational Site 14264, Cincinnati, Ohio
  - Teva Investigational Site 14257, Oklahoma City, Oklahoma
  - Teva Investigational Site 14275, Oklahoma City, Oklahoma
  - Teva Investigational Site 14363, Tulsa, Oklahoma
  - Teva Investigational Site 14364, Philadelphia, Pennsylvania
  - Teva Investigational Site 14374, Bristol, Tennessee
  - Teva Investigational Site 14252, Austin, Texas
  - Teva Investigational Site 14273, Austin, Texas
  - Teva Investigational Site 14274, Bellaire, Texas
  - Teva Investigational Site 14367, Dallas, Texas
  - Teva Investigational Site 14312, Houston, Texas
  - Teva Investigational Site 14366, San Antonio, Texas
  - Teva Investigational Site 14241, San Antonio, Texas
  - Teva Investigational Site 14375, Salt Lake City, Utah
  - Teva Investigational Site 14323, Norfolk, Virginia
  - Teva Investigational Site 14277, Tacoma, Washington
- Canada (4):
  - Teva Investigational Site 11180, Ajax, Ontario
  - Teva Investigational Site 11182, Ottawa, Ontario
  - Teva Investigational Site 11179, Ottawa, Ontario
  - Teva Investigational Site 11181, Montreal, Quebec
- Finland (4):
  - Teva Investigational Site 40053, Helsinki
  - Teva Investigational Site 40049, Kuopio
  - Teva Investigational Site 40054, Oulu
  - Teva Investigational Site 40052, Tampere
- Germany (5):
  - Teva Investigational Site 32728, Bad Homburg
  - Teva Investigational Site 32729, Berlin
  - Teva Investigational Site 32725, Dresden
  - Teva Investigational Site 32724, Essen
  - Teva Investigational Site 32726, Leipzig
- Israel (7):
  - Teva Investigational Site 80170, Be’er Ya‘aqov
  - Teva Investigational Site 80166, Haifa
  - Teva Investigational Site 80168, Holon
  - Teva Investigational Site 80169, Jerusalem
  - Teva Investigational Site 80167, Ramat Gan
  - Teva Investigational Site 80164, Safed
  - Teva Investigational Site 80165, Tel Aviv
- Italy (7):
  - Teva Investigational Site 30230, Florence
  - Teva Investigational Site 30239, Milan
  - Teva Investigational Site 30228, Milan
  - Teva Investigational Site 30226, Milan
  - Teva Investigational Site 30238, Padua
  - Teva Investigational Site 30227, Pavia
  - Teva Investigational Site 30225, Rome
- Netherlands (3):
  - Teva Investigational Site 38138, Doetinchem
  - Teva Investigational Site 38135, Nijmegen
  - Teva Investigational Site 38136, Rotterdam
- Poland (8):
  - Teva Investigational Site 53441, Gdansk
  - Teva Investigational Site 53437, Kielce
  - Teva Investigational Site 53443, Krakow
  - Teva Investigational Site 53452, Krakow
  - Teva Investigational Site 53440, Lublin
  - Teva Investigational Site 53439, Poznan
  - Teva Investigational Site 53451, Poznan
  - Teva Investigational Site 53442, Szczecin
- Spain (6):
  - Teva Investigational Site 31271, Barcelona
  - Teva Investigational Site 31266, Elda
  - Teva Investigational Site 31268, Madrid
  - Teva Investigational Site 31267, Madrid
  - Teva Investigational Site 31270, Valencia
  - Teva Investigational Site 31265, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request

REFERENCES:
- [Derived] Hershey AD, Szperka CL, Barbanti P, Pozo-Rosich P, Bittigau P, Barash S, Bryson J, Kessler Y, Carmeli Schwartz Y, Ramirez Campos V, Ning X. Fremanezumab in Children and Adolescents with Episodic Migraine. N Engl J Med. 2026 Jan 15;394(3):243-252. doi: 10.1056/NEJMoa2504546. PMID 41534042

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 411 participants were screened; of which 235 participants were randomized and included in the analysis.
Groups:
- Placebo: Participants received placebo matched to fremanezumab SC for 3 months (Days 1, 29, and 57).
- Fremanezumab Dose A: Participants weighing <threshold weight received fremanezumab SC at dose A for 3 months (Days 1, 29, and 57).
- Fremanezumab Dose B: Participants weighing ≥threshold weight received fremanezumab SC at dose B for 3 months (Days 1, 29, and 57).
Period: Overall Study
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Started | 112 | 36 | 87
Received at Least 1 Dose of Study Drug | 112 | 36 | 87
Completed | 106 | 33 | 86
Not Completed | 6 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B | Total
Number analyzed (Participants) | 112 | 36 | 87 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.99) | 11.0 (2.27) | 14.2 (2.34) | 13.3 (2.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 16 | 50 | 130
  Male | 48 | 20 | 37 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 8 | 21
  Not Hispanic or Latino | 102 | 31 | 75 | 208
  Unknown or Not Reported | 1 | 1 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 4 | 9
  White | 84 | 28 | 68 | 180
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 24 | 7 | 13 | 44
Number of Migraine Days Per Month [Mean (Standard Deviation); unit: migraine days per month] — A migraine day was defined as a day with either of the following: A day (0:00 to 23:59) with at least 2 hours of headache with ≥2 migraine symptom(s) or day (0:00 to 23:59) demonstrating a headache treated with migraine medications (e.g., non-steroidal anti-inflammatory drugs [NSAIDs], paracetamol etc.). The number of migraine days during baseline was calculated using headache diary data collected in the run-in period and normalized to a 28-day equivalent using formula: (Total migraine days during run-in/Total days with assessments recorded in the diary for the run-in period) × 28.
  migraine days per month | 7.5 (2.84) | 7.6 (2.92) | 7.9 (3.21) | 7.7 (2.99)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Monthly Average Number of Migraine Days During 12-Week Period After the First Dose of Study Drug
Description: A migraine day was defined as a day with any of the following: A day (0:00 to 23:59) with at least 2 hours of headache with ≥2 migraine symptom(s) or day (0:00 to 23:59) demonstrating a headache treated with migraine medications (e.g., non-steroidal anti-inflammatory drugs [NSAIDs], paracetamol etc.), or a headache associated with aura. Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in electronic diary (e-diary) for 12-week period) * 28. Least square (LS) mean was calculated using analysis of covariance (ANCOVA). The full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug and had at least 10 days of diary entries postbaseline for efficacy assessments on primary endpoint. Efficacy analysis was planned to be collected and evaluated combined for both fremanezumab dose treatment groups.
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug and had at least 10 days of diary entries postbaseline for efficacy assessments on the primary endpoint. Efficacy analysis was planned to be evaluated combined for both fremanezumab dose treatment groups.
Measure: Least Squares Mean (Standard Error); unit: days/month
Groups:
- Fremanezumab: Participants received fremanezumab SC for 3 months (Days 1, 29, and 57).
Arm/Group | Placebo | Fremanezumab
Number analyzed (Participants) | 111 | 123
days/month | -1.4 (0.39) | -2.5 (0.38)
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab; Test type: Other; p = 0.0210, ANCOVA; LS mean Difference = -1.0, 95% CI 2-sided [-1.90 to -0.16], Standard Error of Mean 0.44

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. AEs were considered TEAEs if onset occurred on or after the first dose date. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Month 3
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 112 | 36 | 87
Participants | 55 | 20 | 48

3. Secondary Outcome: Number of Participants With Shift From Baseline to Last Assessment in Electrocardiogram (ECG) Findings (Assessed by Investigator)
Description: The number of participants with a shift from Baseline (Normal, Abnormal CS [Clinically Significant], or Abnormal NCS [Not Clinically Significant]) in any of the following ECG parameters is reported by treatment group: Heart rate, PR interval, QRS interval, RR interval, QT interval, QT interval corrected using the Bazett's formula (QTcB), and QT interval corrected using the Fridericia formula (QTcF). Last assessment was defined as the last observed postbaseline interpretation. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline to last assessment (up to Month 3)
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 112 | 36 | 87
Participants
  Normal/Normal | 92 | 32 | 74
  Abnormal NCS/Normal | 13 | 0 | 4
  Abnormal CS/Normal | 0 | 0 | 0
  Normal/Abnormal NCS | 2 | 2 | 6
  Abnormal NCS/Abnormal NCS | 4 | 1 | 3
  Abnormal CS/Abnormal NCS | 0 | 0 | 0
  Normal/Abnormal CS | 0 | 0 | 0
  Abnormal NCS/Abnormal CS | 0 | 0 | 0
  Abnormal CS/Abnormal CS | 0 | 0 | 0
  Missing | 1 | 1 | 0

4. Secondary Outcome: Number of Participants With Shift From Baseline to Last Assessment in ECG Findings (Assessed by Cardiologist)
Description: The number of participants with a shift from Baseline (Normal or Abnormal) in any of the following ECG parameters is reported by treatment group: Heart rate, PR interval, QRS interval, RR interval, QT interval, QTcB, and QTcF. Last assessment was defined as the last observed postbaseline interpretation. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline to last assessment (up to Month 3)
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 112 | 36 | 87
Participants
  Normal/Normal | 88 | 29 | 72
  Abnormal/Normal | 14 | 0 | 5
  Normal/Abnormal | 2 | 4 | 4
  Abnormal/Abnormal | 6 | 2 | 6
  Missing | 2 | 1 | 0

5. Secondary Outcome: Number of Participants With Any One or More Potentially Clinically Significant Vital Signs Abnormalities
Description: Potentially clinically significant abnormal vital signs findings included any one of the following: Pulse rate ≥120 beats per minute (bpm) and increase from baseline of ≥15 bpm, or ≤50 bpm and decrease from baseline of ≥15 bpm; Systolic blood pressure ≤85 millimeters of mercury (mmHg) and decrease from baseline of ≥20 mmHg; Diastolic blood pressure ≥100 mmHg and increase from baseline of ≥15 mmHg; Respiratory rate <15 breaths/minute. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Month 3
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' = participants with at least one Baseline and post-baseline vital sign assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 112 | 35 | 87
Participants | 14 | 3 | 5

6. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory (Serum Chemistry, Hematology, Coagulation, and Urinalysis) Results
Description: Serum chemistry tests with potentially clinically significant abnormal findings included: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) both ≥2*upper limit of normal (ULN); and bilirubin ≥34.2 micromole/liter (umol/L). Hematology tests with potentially clinically significant abnormal findings included: hemoglobin ≤100 grams (g)/L, leukocytes ≤3*10^9 cells/L, neutrophils ≤1*10^9 cells/L, eosinophils/leukocytes ≥10%, and platelets ≥700*10^9 cells/L or ≤75*10^9 cells/L. Coagulation parameter test with potentially clinically significant abnormal findings included: prothrombin international normalized ratio (INR) >1.5. Urinalysis laboratory tests with potentially clinically significant abnormal findings included: urine protein ≥2 units (U) increase from baseline. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Month 3
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' and 'Number analyzed'= participants with at least one Baseline and post-baseline assessment of the specified laboratory parameters.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 111 | 35 | 87
Participants
  With at least 1 serum chemistry abnormality | 2 | 1 | 3
  With at least 1 hematology abnormality: number analyzed (Participants) | 110 | 34 | 87
  With at least 1 hematology abnormality | 6 | 2 | 3
  With at least 1 coagulation abnormality: number analyzed (Participants) | 110 | 35 | 87
  With at least 1 coagulation abnormality | 3 | 0 | 1
  With at least 1 urinalysis abnormality | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings as Identified by the Investigator
Description: A complete physical examination included the following organ systems: general appearance; head, eyes, ears, nose, and throat (HEENT); chest and lungs; heart; abdomen; musculoskeletal; skin; lymph nodes; and neurological. Only the organ systems with abnormal physical findings in at least one treatment group have been reported. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Month 3
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' = participants with at least one Baseline and post-baseline physical examination.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 109 | 34 | 87
Participants
  General Appearance | 0 | 0 | 1
  HEENT | 1 | 0 | 1
  Musculoskeletal | 2 | 0 | 1
  Skin | 5 | 1 | 2
  Neurological | 1 | 0 | 0
  Extremities/Back | 0 | 0 | 1

8. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation was defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent.
Time Frame: Baseline and Month 3
Population: The ITT analysis set included all randomized participants. Here, 'Overall number of participants analyzed' = participants with both Baseline and Month 3 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 105 | 33 | 86
Participants
  Baseline | 0 | 1 | 0
  Month 3 | 1 | 0 | 0

9. Secondary Outcome: Mean Change From Baseline in Monthly Average Number of Headache Days of at Least Moderate Severity During 12-Week Period After the First Dose of Study Drug
Description: A headache day of at least moderate severity was defined as a calendar day (00:00 to 23:59) where the participant reported either of the following: A day with headache pain that lasted ≥2 hours with a peak severity of at least moderate severity or a day where the participant used acute medication (triptans, ergots, NSAIDs or paracetamol) to treat a headache of any severity or duration. Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in e-diary for 12-week period) * 28. LS mean was calculated using ANCOVA.
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: The FAS included all randomized participants who received at least 1 dose of study drug and had at least 10 days of diary entries postbaseline for efficacy assessments on the primary endpoint. Efficacy analysis was planned to be evaluated combined for both fremanezumab dose treatment groups.
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab
Number analyzed (Participants) | 111 | 123
days/month | -1.5 (0.42) | -2.6 (0.40)

10. Secondary Outcome: Number of Participants Reaching at Least 50% Reduction in the Monthly Average Number of Migraine Days During the 12-week Period After the First Dose of Study Drug
Description: A migraine day was defined as a calendar day where the participant reported either of the following: A calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache that was accompanied by ≥1 migraine symptom(s) or a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine specific medications (NSAIDs, paracetamol or triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in e-diary for 12-week period) * 28.
Time Frame: Baseline (Day -28 to Day -1) up to Week 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab
Number analyzed (Participants) | 111 | 123
Participants | 30 | 58

11. Secondary Outcome: Mean Change From Baseline in Monthly Average Number of Days of Use of Any Acute Headache Medications During 12-Week Period After the First Dose of Study Drug
Description: Participants recorded any headache medications (name of drug, number of tablets/capsules, and the dose in milligrams per tablet/capsule) taken each day in their electronic headache diary device. Acute headache medication included triptans and ergot compounds, NSAIDs or paracetamol. Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in e-diary for 12-week period) * 28. LS mean was calculated using ANCOVA.
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab
Number analyzed (Participants) | 111 | 123
days/month | -1.0 (0.30) | -2.1 (0.29)

12. Secondary Outcome: Mean Change From Baseline in Migraine-related Disability Score at Week 12, as Measured by the Pediatric Migraine Disability Assessment (PedMIDAS) Questionnaire
Description: The PedMIDAS is a scale developed to assess headache-related disability which can be self-administered by the participant or administered by a caregiver. It has been validated in participants aged 4 to 18 years and includes 3 subscales: the impact of headache on school performance (range of scores 0-92), disability at home (range of scores 0-92), social/sport functioning (range of scores 0-92). The subscales are added to get the total score with a range 0 to 276. The total score was used for grading of disability, with 4 score categories of 0 to 10, 11 to 30, 31 to 50, and 51-276 interpreted as disability grades 1 (little or no disability), 2 (mild disability), 3 (moderate disability), and 4 (severe disability), respectively. Higher total scores indicated severe disability. LS mean was calculated using ANCOVA. The change from baseline score is reported with a range of -276 to 276 with higher scores indicating more severe disability.
Time Frame: Baseline, Week 12
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fremanezumab
Number analyzed (Participants) | 111 | 123
units on a scale | -15.3 (3.37) | -21.6 (3.29)

13. Secondary Outcome: Mean Change From Baseline in Quality of Life at Week 12, as Measured by Pediatric Quality of Life Inventory (PedsQL) Questionnaire
Description: PedsQL 4.0 is a brief 23-item health-related quality of life (QoL) instrument that evaluates QoL in 4 areas of functioning: physical, emotional, social, and school functioning. For child and adolescent self-report (8 - 18 years) and parent report forms, respondents used a 5-point Likert scale to rate item severity (0=never a problem;1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem). For younger children (5 - 7 years), a simplified 3-point Likert scale, anchored with a happy and a sad face, was used (0=not at all a problem; 2=sometimes a problem; 4=a lot of a problem). PedsQL yields a total QoL score and 2 summary scores: Physical Health Summary Score and Psychosocial Health Summary Score. To obtain scores, items were reverse scored, transformed to a 0 through 100 scale (0=100, 1=75, 2=50, 3=25, 4=0), and averaged; total scores near 0 indicated lower QoL, while scores approaching 100 indicated higher QoL. LS mean was calculated using ANCOVA.
Time Frame: Baseline, Week 12
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Fremanezumab
Number analyzed (Participants) | 111 | 123
units on a scale
  Child-Physical Health Summary Score | 8.3 (1.61) | 7.8 (1.57)
  Child-Psychosocial Health Summary Score | 5.3 (1.38) | 4.7 (1.35)
  Child-Total Scale Score | 6.2 (1.37) | 5.7 (1.33)
  Parent-Physical Health Summary Score | 7.3 (2.69) | 7.3 (2.35)
  Parent-Psychosocial Health Summary Score | 6.8 (2.28) | 4.3 (1.96)
  Parent-Total Scale Score | 7.2 (2.28) | 5.2 (1.97)

14. Secondary Outcome: Number of Participants Developing Anti-drug Antibodies (ADAs) Throughout the Study
Description: Number of participants who developed ADAs were reported.
Time Frame: Baseline up to Month 3
Population: The FAS included all randomized participants who received at least 1 dose of study drug and had at least 10 days of diary entries postbaseline for efficacy assessments on the primary endpoint. Here, 'Overall number of participants analyzed' = Participants who had Baseline and at least 1 postbaseline ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 35 | 87
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Month 3
Description: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/36 | 0/87
Serious Adverse Events (participants affected / at risk) | 3/112 | 1/36 | 1/87
Other Adverse Events (participants affected / at risk) | 26/112 | 8/36 | 29/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=112) | Fremanezumab Dose A (N=36) | Fremanezumab Dose B (N=87)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=112) | Fremanezumab Dose A (N=36) | Fremanezumab Dose B (N=87)
Injection site erythema (General disorders) | 6 (9) | 1 (2) | 11 (18)
Injection site pain (General disorders) | 6 (10) | 0 (0) | 6 (9)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 5 (6)
Vaccination site pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 2 (2) | 5 (5)
Nasopharyngitis (Infections and infestations) | 8 (10) | 3 (4) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 2 (2) | 4 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 2 (3) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2023-09-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT04458857/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT04458857/SAP_002.pdf